CLINICAL TRIAL: NCT02976272
Title: Assessment of Sensory Disorders Associated With Peripheral Neuropathy Induced by Bortezomib: Prospective Comparative Study
Brief Title: Neurotoxic Effect of Bortezomib Treatment in Patient With Myeloma Multiple
Acronym: SENSIB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Laboratoires Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: CHU-0291; 2015-A01172-47 (Other: 2015-A01172-47)
Record Dates: First submitted 2016-11-18; First posted 2016-11-29 (Estimated); Last update posted 2019-07-01 (Actual); Status verified 2016-11

CONDITIONS: Multiple Myeloma; Bortezomib Regimen; Adult
Keywords: Bortezomib regimen; patients with multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- patients with myeloma multiple
  Interventions: Other: bortezomib

INTERVENTIONS:
Other: bortezomib

SUMMARY:
Chemotherapy-induced peripheral neuropathies (CIPN) remain a problem in oncology because no "gold standard" treatment exists to prevent or treat the CIPN. Therefore, oncologists reduce or stop the chemotherapy doses to limit degradation of the quality of life of patients with CIPN. Bortezomib is relatively understudied while neurotoxicity remains a limiting factor for treatment. Since 2012, the FDA and the EMA validated by the administration of bortezomib subcutaneously (SC) instead of intravenous (IV) in order to limit neurotoxicity.

However, a retrospective study reported that the prevalence of neuropathy induced by bortezomib after SC administration remains high and equivalent to IV route. No studies have quantitatively and qualitatively evaluated the sensory disorders in peripheral neuropathies induced by bortezomib after SC administration. On the other hand, the QLQ-CIPN20 questionnaire (EORTC) evaluating the intensity of sensory, motor and autonomic disorders associated with CIPN has never been tested in this population. The objective of this study is twofold: (i) psychophysical evaluation of neuropathic disorders by studying the thermal and vibratory detection thresholds and thermal nociceptive thresholds and (ii) quantitative and qualitative assessment of neuropathic disorders by the QLQ-CIPN20 and related comorbidities in a population of neuropathic patients treated with bortezomib (n = 15), compared to control patients treated with bortezomib but non-neuropathic (n = 45).

DETAILED DESCRIPTION:
Peripheral neuropathies induced by cancer chemotherapy (CIPN) remain a problem in oncology. These CIPN are induced by certain classes of chemotherapy such as taxanes (paclitaxel and docetaxel), platinum salts (cisplatin and oxaliplatin), alkaloids of the Madagascar periwinkle (vincristine), bortezomib, thalidomide and eribulin. These CIPN is essentially resulting in sensory disturbances such as paresthesia, dysesthesia or numbness. Unfortunately, no treatment can be offered as "gold standard" for preventing or treating the CIPN. Therefore, oncologists reduce or stop doses of chemotherapy because patients suffering from CIPN have a marked deterioration in their quality of life and suffer from comorbidities such as anxiety, depression and sleep disorders.

Among chemotherapy, bortezomib remains relatively understudied in terms of pathophysiology, compared to the platinum salts or taxanes, whereas the neurotoxicity of bortezomib remains a limiting factor for treatment. Currently, bortezomib is indicated for the treatment in 1st line of multiple myeloma in the following protocols:

* Patients <65 years: Protocol VTD: Velcade (bortezomib), thalidomide, dexamethasone + autologous transplant
* Patients> 65: Protocol MPV: Melphalan, Prednisone, Velcade. Or Protocol VD: Velcade, dexamethasone Since 2012, the FDA and the EMA have validated the subcutaneous administration of bortezomib instead of intravenously, in order to limit the adverse effects of bortezomib, including neurotoxicity. Indeed, a large study reported that the subcutaneous bortezomib allowed to keep the same therapeutic efficacy while improving the safety profile and in particular by limiting peripheral neuropathies (CIPN any grade: 38% vs 53%, grade ≥2: 24% vs 41%, grade ≥3 6% vs 16%). However, a recent retrospective study reported that the prevalence of peripheral neuropathies induced by bortezomib after subcutaneous administration remain relatively high: CIPN any grade: 41%, grade ≥2: 18% grade ≥3: 4 %, and especially that this prevalence of CIPN is no different between subcutaneous and intravenous route.

Bortezomib is administered subcutaneously to limit the appearance of neuropathic disorders and no study has evaluated quantitatively and qualitatively (QST) the sensory disorders in patients with peripheral neuropathies induced by bortezomib after subcutaneous administration. On the other hand, a measurement tool like the QLQ-CIPN20 questionnaire (EORTC) evaluating the intensity of sensory, motor and autonomic disorders associated with CIPN has never been tested in this patient population. While the questionnaire is presented as the most appropriate tool in the evaluation of CIPN.

Thus, the exploration of peripheral neuropathies induced by bortezomib after subcutaneous administration through QST (thermal) and QLQ-CIPN20 questionnaire would complement the clinical knowledge of the CIPN. This knowledge will be essential to propose and test new strategies for treatment and prevention of peripheral neuropathies induced by bortezomib.

The objective of this study is twofold: (i) psychophysical evaluation of neuropathic disorders by studying the QST (thermal and vibratory sensory thresholds, thermal nociceptive thresholds) and (ii) quantitative and qualitative assessment of neuropathic disorders by the QLQ -CIPN20 questionnaire (EORTC) and associated comorbidities in patients treated with bortezomib (subcutaneous administration).

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma diagnosis.
* Patient undergoing or who received bortezomib-based chemotherapy in first-line (VTD protocol, MPV or VD).

Case Group: peripheral sensory neuropathy

* Neuropathy ≥ grade 2 (grade 2-3) from NCI-CTCAE

Control group: asymptomatic

* Neuropathy of grade <2 (grade 0-1) from NCI-CTCAE

Exclusion Criteria:

* Age <18 years.
* Treatment history by neurotoxic chemotherapy (taxanes, platinum salts, bortezomib, thalidomide, eribulin) before the current treatment.
* Existing treatment: opioids, tricyclic antidepressants, pregabalin, gabapentin, duloxetine or AEDs.
* Drinking: Male > 3 and Woman > 2 units per day.
* Peripheral neuropathies history or known neuropathic pain
* Progressive neurological disease.
* Patient enrolled in a clinical study evaluating a preventive or curative treatment of chemotherapy-induced peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with myeloma multiple
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-06-07 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Thermal sensory thresholds of sensitivity to hot measured using a thermode (Medoc TSA-II Abioz Technologies) | at day 1
Sensory thresholds of patients will be measured using a thermode (Medoc TSA-II Abioz Technologies) | at day 1
Thermal sensory thresholds will be reviewed at the thenar eminence of 2 hands | at day 1

SECONDARY OUTCOMES:
Sensitivity to heat, cold and vibration (will be measured using a thermode) | at day 1
Pain induced by hot and cold (will be measured using a thermode) | at day 1
Neuropathic symptoms (DN4 questionnaires) | at day 1
Neuropathic symptoms (QLQ CIPN20 NPSI questionnaires) | at day 1
Neuropathic pain (NRS) measured using a thermode (Medoc TSA-II Abioz Technologies) | at day 1
Quality of life (QLQ-C30 questionnaires) | at day 1
Quality of life (QLQ-MY20 questionnaires) | at day 1
Depression (HADS questionnaire) | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Carine CHALETEIX, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France